CLINICAL TRIAL: NCT02465398
Title: Anatomical Shoulder™ Fracture Post-Market Surveillance Study
Brief Title: Anatomical Shoulder™ Fracture PMCF Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-U03
Record Dates: First submitted 2015-06-04; First posted 2015-06-08 (Estimated); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-02

CONDITIONS: Fracture
Keywords: Fracture shoulder arthroplasty; Three or four part fracture; Hemiarthroplasty; Multi-center; Europe; Non-controlled; Anatomical reconstruction; Proximal
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fracture device (Other): Patient were treated with an Anatomical Shoulder Fracture device.
  Interventions: Procedure: Fracture Shoulder Arthroplasty

INTERVENTIONS:
Procedure: Fracture Shoulder Arthroplasty — Implantation of the Anatomical Shoulder Fracture System

SUMMARY:
The purpose of this study is to obtain outcomes data on the Anatomical Shoulder Fracture System by analysis of standard scoring systems and radiographs.

Outcome data will be collected using the following standard scoring systems:

- Constant and Murley Score

DETAILED DESCRIPTION:
This is a multi-centre, non-comparative, prospective post-market surveillance study involving surgeons skilled in shoulder replacement surgery. Each case enrolled will receive an Anatomical Shoulder Fracture implant. All system components are CE (Conformité Européenne)-marked and commercially available. Patients will be selected according to the subject selection criteria.

All patients will undergo pe-operative, intra-operative and post-operative physical examination, radiographic evaluation according to the hospital's routine procedure and collection of quality of life metrics. Follow-up evaluations are to be conducted at 6-12 weeks (x-rays only), at 6 months and annually thereafter for a minimum period of 5 years post hospital discharge. Follow-up evaluation at 10 years post hospital discharge is optional.

ELIGIBILITY:
Inclusion Criteria:

* Age - 18 years minimum.
* Sex - male and female.
* General Health - the patient should be able to undergo surgery and participate in a follow-up program based upon physical examination and medical history.
* Informed Consent - patient or patient's legal representative has signed a 'Patient Informed Consent form'.
* Indications - Diagnosis of trauma in the affected joint with the indication for shoulder hemiarthroplasty.

Exclusion Criteria:

* Patient is skeletally immature.
* Patient is pregnant.
* Patient is unwilling or unable to cooperate in a follow-up program.
* Patient is planned for a bilateral shoulder replacement.
* Patient shows one or more of the following medical conditions:

  * Pathological Fracture
  * Active Infection
* Patient requires one or more of the following medical interventions:

  * Revision surgery (non-union)
  * Inverse fracture prosthesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-07-05 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2024-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Goff, PhD, Study Chair — Zimmer Biomet, Jr. Clinical Project Lead
Locations (3):
- Klinikum Augsburg, Augsburg, Germany
- Uniklinik Balgrist, Zurich, Switzerland
- The Pennine Acute Hospital NHS Trust, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Implants
Period: Overall Study
Arm/Group | Fracture Device
Started | 52; 52 Implants (52 enrolled, 51 participants received study device)
Completed | 22; 22 Implants (5-year data of 22 were available for analysis.)
Not Completed | 30; 30 Implants
Not completed — Death | 7
Not completed — Revision | 7
Not completed — did not receive study device | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 14

BASELINE CHARACTERISTICS:
Population: 52 subjects enrolled, 51 subjects operated.
Arm/Group | Fracture Device
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 50
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 19
  Switzerland | 24
  Germany | 8
BMI [Mean (Standard Deviation); unit: kg/m2] | 28.4 (8.9)
Height [Mean (Standard Deviation); unit: cm] | 167.6 (10.1)
Weight [Mean (Standard Deviation); unit: kg] | 79.5 (24.0)

OUTCOME MEASURES:

1. Primary Outcome: Functional Performance
Description: Constant & Murley Score. This evaluates clinical parameters such as range of motion, power, level of pain and functional ability. The score ranges from 0 - 100 with a higher score representing a better outcome.
Time Frame: 5 years
Population: 22 participants with Constant & Murley Score between baseline and 5 years follow-up available.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Implants
Arm/Group | Fracture Device
Number analyzed (Participants) | 22
Number analyzed (Implants) | 22
score on a scale | 57.7 (13.2)

ADVERSE EVENTS:
Time Frame: AE data was collected over the entire study from surgery date until an average of 5 years
Description: Seriousness of the Adverse Events were not assessed. Therefore, all Adverse Events are listed in the Serious Adverse Events table
Arm/Group | Fracture Device
All-Cause Mortality (participants affected / at risk) | 7/52
Serious Adverse Events (participants affected / at risk) | 20/52
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fracture Device (N=52)
Death due to unrelated reasons (General disorders) | 7 (7)
Revision: conversion to reverse prosthesis (Surgical and medical procedures) | 6 (6)
Revision: conversion to reverse prosthesis (Surgical and medical procedures) | 1 (1)
Frozen Shoulder (Musculoskeletal and connective tissue disorders) | 3 (3)
Intraoperative fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Nerve deficit (Nervous system disorders) | 1 (1)
Subluxation (Musculoskeletal and connective tissue disorders) | 1 (1)
Heterotopic ossification (Musculoskeletal and connective tissue disorders) | 2 (2)
Other, not shoulder related complications (Musculoskeletal and connective tissue disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-08-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT02465398/Prot_SAP_000.pdf